CLINICAL TRIAL: NCT02063854
Title: A Phase 2/3, Multicenter, Randomized, Double-blind, Parallel Group Comparative Study to Evaluate the Efficacy and Safety of Once-monthly Oral Administration of NE-58095DR Tablet (25 mg or 37.5 mg) Versus Once-daily Oral Administration of NE-58095IR Tablet (2.5 mg) for the Treatment of Involutional Osteoporosis
Brief Title: A Phase II/III, Double-blind, Parallel Group Comparative Study of Oral Administration of NE-58095 Tablets
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: EA Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCT-401; JapicCTI-142440 (Registry Identifier: JapicCTI); U1111-1153-0440 (Registry Identifier: WHO); NE-58095DR/CCT-401 (Other: Takeda ID); NCT02066376 (obsolete NCT alias)
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Involutional Osteoporosis
Keywords: Drug Therapy
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- NE-58095 IR 2.5 mg Once Daily on Awakening (Active Comparator): NE-58095 immediate release (IR) 2.5 mg tablet, orally, once, daily, at time of wakening + NE-58095 delayed release (DR) placebo-matching tablet, orally, once, monthly, at time of wakening + NE-58095 DR placebo-matching tablet, orally, once, monthly, following breakfast + NE-58095 DR placebo-matching tablet, orally, once, monthly, 30 minutes after breakfast, for up to 12 months. Calcium lactate hydrate 195 mg, once, daily, after dinner was taken as a background medication.
  Interventions: Drug: NE-58095 IR; Drug: NE-58095 DR Placebo
- NE-58095 DR 25 mg Once Monthly on Awakening (Experimental): NE-58095 DR 25 mg tablet, orally, once, monthly, at time of wakening + NE-58095 DR placebo-matching tablet, orally, once, monthly, following breakfast + NE-58095 DR placebo-matching tablet, orally, once, monthly, 30 minutes after breakfast + NE-58095 IR placebo-matching tablet, orally, once, daily, at time of wakening, for up to 12 months. Calcium lactate hydrate 195 mg, once, daily, after dinner was taken as a background medication.
  Interventions: Drug: NE-58095 IR Placebo; Drug: NE-58095 DR; Drug: NE-58095 DR Placebo
- NE-58095 DR 25 mg Once Monthly Following Breakfast (Experimental): NE-58095 DR 25 mg tablet, orally, once, monthly, following breakfast + NE-58095 DR placebo-matching tablet, orally, once, monthly, 30 minutes after breakfast + NE-58095 DR placebo-matching tablet, orally, once, monthly, at time of wakening + NE-58095 IR placebo-matching tablet, orally, once, daily, at time of wakening, for up to 12 months. Calcium lactate hydrate 195 mg, once, daily, after dinner was taken as a background medication.
  Interventions: Drug: NE-58095 IR Placebo; Drug: NE-58095 DR; Drug: NE-58095 DR Placebo
- NE-58095 DR 25 mg Once Monthly 30 Min. After Breakfast (Experimental): NE-58095 DR 25 mg tablet, orally, once, monthly, 30 minutes after breakfast + NE-58095 DR placebo-matching tablet, orally, once, monthly, following breakfast + NE-58095 DR placebo-matching tablet, orally, once, monthly, at time of wakening + NE-58095 IR placebo-matching tablet, orally, once, daily, at time of wakening, for up to 12 months. Calcium lactate hydrate 195 mg, once, daily, after dinner was taken as a background medication.
  Interventions: Drug: NE-58095 IR Placebo; Drug: NE-58095 DR; Drug: NE-58095 DR Placebo
- NE-58095 DR 37.5 mg Once Monthly on Awakening (Experimental): NE-58095 DR 37.5 mg tablet, orally, once, monthly, at time of wakening + NE-58095 DR placebo-matching tablet, orally, once, monthly, following breakfast + NE-58095 DR placebo-matching tablet, orally, once, monthly, 30 minutes after breakfast + NE-58095 IR placebo-matching tablet, orally, once, daily, at time of wakening, for up to 12 months. Calcium lactate hydrate 195 mg, once, daily, after dinner was taken as a background medication.
  Interventions: Drug: NE-58095 IR Placebo; Drug: NE-58095 DR; Drug: NE-58095 DR Placebo
- NE-58095 DR 37.5 mg Once Monthly Following Breakfast (Experimental): NE-58095 DR 37.5 mg tablet, orally, once, monthly, following breakfast + NE-58095 DR placebo-matching tablet, orally, once, monthly, 30 minutes after breakfast + NE-58095 DR placebo-matching tablet, orally, once, monthly, at time of wakening + NE-58095 IR placebo-matching tablet, orally, once, daily, at time of wakening, for up to 12 months. Calcium lactate hydrate 195 mg, once, daily, after dinner was taken as a background medication.
  Interventions: Drug: NE-58095 IR Placebo; Drug: NE-58095 DR; Drug: NE-58095 DR Placebo
- NE-58095 DR 37.5 mg Once Monthly 30 Min. After Breakfast (Experimental): NE-58095 DR 37.5 mg tablet, orally, once, monthly, 30 minutes after breakfast + NE-58095 DR placebo-matching tablet, orally, once, monthly, following breakfast + NE-58095 DR placebo-matching tablet, orally, once, monthly, at time of wakening + NE-58095 IR placebo-matching tablet, orally, once, daily, at time of wakening, for up to 12 months. Calcium lactate hydrate 195 mg, once, daily, after dinner was taken as a background medication.
  Interventions: Drug: NE-58095 IR Placebo; Drug: NE-58095 DR; Drug: NE-58095 DR Placebo

INTERVENTIONS:
Drug: NE-58095 IR — NE-58095 IR tablets
  Arms: NE-58095 IR 2.5 mg Once Daily on Awakening
Drug: NE-58095 IR Placebo — NE-58095 IR placebo-matching tablets
  Arms: NE-58095 DR 25 mg Once Monthly 30 Min. After Breakfast; NE-58095 DR 25 mg Once Monthly Following Breakfast; NE-58095 DR 25 mg Once Monthly on Awakening; NE-58095 DR 37.5 mg Once Monthly 30 Min. After Breakfast; NE-58095 DR 37.5 mg Once Monthly Following Breakfast; NE-58095 DR 37.5 mg Once Monthly on Awakening
Drug: NE-58095 DR — NE-58095 DR tablets
  Arms: NE-58095 DR 25 mg Once Monthly 30 Min. After Breakfast; NE-58095 DR 25 mg Once Monthly Following Breakfast; NE-58095 DR 25 mg Once Monthly on Awakening; NE-58095 DR 37.5 mg Once Monthly 30 Min. After Breakfast; NE-58095 DR 37.5 mg Once Monthly Following Breakfast; NE-58095 DR 37.5 mg Once Monthly on Awakening
Drug: NE-58095 DR Placebo — NE-58095 DR placebo-matching tablets

SUMMARY:
The present phase II/III, multicenter, randomized, double-blind, parallel group comparative study is designed to evaluate the efficacy and safety of once-monthly oral administration of NE-58095 delayed release (DR) tablets for 12 months in participants with involutional osteoporosis. For this study, participants receiving oral NE-58095 immediate release (IR) 2.5 mg tablets once daily for 12 months are set as the control group.

DETAILED DESCRIPTION:
The primary objective of the present study is to verify the non-inferiority of once-monthly oral administration of NE-58095 DR tablets for 12 months to once-daily oral administration of NE-58095 IR 2.5 mg tablets for 12 months, in terms of efficacy in participants with involutional osteoporosis.

Secondary objectives of the present study are as follows: to compare the safety of once-monthly oral administration of NE-58095 DR tablets for 12 months with the safety of once-daily oral administration of NE-58095 IR tablets (at 2.5 mg) for 12 months in participants with involutional osteoporosis at time of wakening.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of involutional osteoporosis
2. Male or female outpatients (including patients admitted to the hospital for tests) aged ≥ 50 years at the time of consent
3. Women for whom at least 2 years have passed since the last natural menstruation

Exclusion Criteria:

1. Patients with secondary osteoporosis
2. Patients with diseases (other than secondary osteoporosis) that present with decreased bone mass
3. Patients with findings that affects the measurement of mean bone mineral density of the lumbar spine by dual-energy X-ray absorptiometry (DXA)
4. Patients with a history of radiotherapy to the lumbar spine or the pelvis
5. Patients who are planning to receive surgical dental procedures such as tooth extraction (including dental implant treatment) during the treatment period
6. Patients with a history of treatment with any anti-receptor activator of nuclear factor-κB ligand (RANKL) monoclonal antibodies or parathyroid hormone products within 1 year before the start of the treatment period
7. Patients with a history of treatment with any bisphosphonate products within 24 weeks before the start of the treatment period
8. Patients who have received any drugs that affect bone metabolism within 8 weeks before the start of the treatment period
9. Patients with disorders such as esophagitis, peptic ulcer (e.g., esophageal ulcer, gastric ulcer, and duodenal ulcer), or gastrointestinal bleeding
10. Patients with disorders that delay esophageal emptying (e.g., dysphagia, esophagostenosis, or achalasia of the esophagus)
11. Patients with hypocalcemia
12. Patients with hypercalcemia
13. Patients with a diagnosis of renal calculus
14. Patients with serious renal, hepatic, or cardiac disease
15. Patients who have received surgical dental procedures, such as a tooth extraction (including dental implant treatment), but whose dental problems remain unresolved at the start of the treatment period.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 871 (Actual)
Dates: Start 2014-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (25):
- Japan (25):
  - Nagoya, Aichi-ken
  - Chiba, Chiba
  - Narashino-shi, Chiba
  - Fukuoka, Fukuoka
  - Kitakyushu-shi, Fukuoka
  - Onga-gun, Fukuoka
  - Ebetsu-shi, Hokkaido
  - Sapporo, Hokkaido
  - Kako-gun, Hyōgo
  - Morioka, Iwate
  - Atsugi-shi, Kanagawa
  - Kawasaki-shi, Kanagawa
  - Yokohama, Kanagawa
  - Zushi-shi, Kanagawa
  - Kumamoto, Kumamoto
  - Tamana-shi, Kumamoto
  - Sendai, Miyagi
  - Tagajō-shi, Miyagi
  - Miyazaki, Miyazaki
  - Saito-shi, Miyazaki
  - Higashi Osaka-shi, Osaka
  - Saitama-shi, Saitama
  - Daito-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Wakayama, Wakayama

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 67 investigative sites in Japan from 21 February 2014 to 19 November 2015.
Pre-assignment Details: Participants with a diagnosis of involutional osteoporosis were randomized at a ratio of 3:1:3:1:1:3:1 into 1 of 7 treatment groups: once-daily NE-58095 2.5 mg immediate release (IR) or once-monthly NE-58095 25 mg or 37.5 mg delayed release (DR) on awakening, after breakfast or 30 minutes following breakfast.
Period: Overall Study
Arm/Group | NE-58095 IR 2.5 mg Once Daily on Awakening | NE-58095 DR 25 mg Once Monthly on Awakening | NE-58095 DR 25 mg Once Monthly Following Breakfast | NE-58095 DR 25 mg Once Monthly 30 Min. After Breakfast | NE-58095 DR 37.5 mg Once Monthly on Awakening | NE-58095 DR 37.5 mg Once Monthly Following Breakfast | NE-58095 DR 37.5 mg Once Monthly 30 Min. After Breakfast
Started | 199 | 66 | 206 | 68 | 65 | 201 | 66
Full Analysis Set: Received Study Drug | 199 | 66 | 206 | 68 | 65 | 200 | 66
Completed | 178 | 54 | 176 | 58 | 54 | 170 | 60
Not Completed | 21 | 12 | 30 | 10 | 11 | 31 | 6
Not completed — Pretreatment Event/Adverse Event | 13 | 10 | 13 | 8 | 7 | 18 | 4
Not completed — Major Protocol Deviation | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Voluntary Withdrawal | 2 | 0 | 8 | 1 | 3 | 6 | 1
Not completed — Surgical Dental Work Performed/Planned | 5 | 2 | 6 | 1 | 1 | 6 | 1
Not completed — Reason Not Specified | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Did Not Receive Study Drug | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized set included all participants who were randomized to the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | NE-58095 IR 2.5 mg Once Daily on Awakening | NE-58095 DR 25 mg Once Monthly on Awakening | NE-58095 DR 25 mg Once Monthly Following Breakfast | NE-58095 DR 25 mg Once Monthly 30 Min. After Breakfast | NE-58095 DR 37.5 mg Once Monthly on Awakening | NE-58095 DR 37.5 mg Once Monthly Following Breakfast | NE-58095 DR 37.5 mg Once Monthly 30 Min. After Breakfast | Total
Number analyzed (Participants) | 199 | 66 | 206 | 68 | 65 | 201 | 66 | 871
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (7.32) | 69.0 (8.18) | 68.2 (7.68) | 68.4 (7.24) | 69.0 (6.98) | 69.6 (7.19) | 69.8 (7.87) | 68.9 (7.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 64 | 203 | 66 | 63 | 198 | 63 | 847
  Male | 9 | 2 | 3 | 2 | 2 | 3 | 3 | 24
Region of Enrollment [Number; unit: participants]
  Japan | 199 | 66 | 206 | 68 | 65 | 201 | 66 | 871
Height [Mean (Standard Deviation); unit: cm] | 152.1 (6.59) | 151.0 (6.64) | 151.9 (6.11) | 152.5 (5.49) | 153.5 (5.13) | 151.3 (5.20) | 151.9 (6.47) | 151.9 (6.00)
Weight [Mean (Standard Deviation); unit: kg] — Data was available for 199, 66, 206, 68, 65, 200 and 66 participants in each treatment arm, respectively.
  kg | 50.52 (7.975) | 49.98 (6.720) | 50.20 (7.231) | 50.97 (8.736) | 51.26 (7.473) | 50.36 (7.383) | 50.51 (7.427) | 50.46 (7.544)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Data was available for 199, 66, 206, 68, 65, 200 and 66 participants in each treatment arm, respectively.
  kg/m^2 | 21.82 (3.009) | 21.93 (2.830) | 21.75 (2.926) | 21.97 (3.875) | 21.79 (3.289) | 22.00 (3.105) | 21.90 (3.071) | 21.87 (3.092)
Smoking Classification [Number; unit: participants]
  Never smoked | 167 | 55 | 178 | 53 | 54 | 168 | 58 | 733
  Current smoker | 10 | 4 | 11 | 3 | 3 | 7 | 3 | 41
  Ex-smoker | 22 | 7 | 17 | 12 | 8 | 26 | 5 | 97
Menopausal Status [Number; unit: participants] — Female participants only (N=190, 64, 203, 66, 63, 198, 63).
  participants
    Natural Menopause | 170 | 58 | 179 | 60 | 53 | 180 | 59 | 759
    Artificial Menopause | 20 | 6 | 24 | 6 | 10 | 18 | 4 | 88
Number of Years After Menopause, Categorical [Number; unit: participants] — Female participants only (N=190, 64, 203, 66, 63, 198, 63).
  participants
    Min - ≤5 years | 6 | 5 | 7 | 4 | 3 | 4 | 2 | 31
    6 - ≤10 years | 23 | 1 | 28 | 4 | 8 | 22 | 6 | 92
    11 - ≤20 years | 59 | 21 | 71 | 29 | 20 | 61 | 20 | 281
    21 - ≤30 years | 55 | 19 | 42 | 12 | 19 | 58 | 19 | 224
    ≥31 years | 9 | 6 | 11 | 7 | 4 | 17 | 4 | 58
    Unknown, But >2 years | 38 | 12 | 44 | 10 | 9 | 36 | 12 | 161
Number of Years After Menopause [Mean (Standard Deviation); unit: years] — Data was available for 152, 52, 159, 56, 54, 162 and 51 female participants in each treatment arm, respectively.
  years | 18.6 (7.81) | 20.2 (8.72) | 17.2 (8.44) | 18.3 (8.28) | 19.2 (8.36) | 19.5 (8.41) | 20.1 (7.84) | 18.7 (8.28)
History of Bisphosphonate Administration [Number; unit: participants]
  Yes | 19 | 6 | 24 | 8 | 9 | 26 | 6 | 98
  No | 180 | 60 | 182 | 60 | 56 | 175 | 60 | 773
Timing of Initial Delayed Release (DR) Tablet Administration on Awakening [Number; unit: participants] — Data was available for 199, 66, 206, 68, 65, 200 and 66 participants in each treatment arm, respectively.
  participants
    Less than 30 Minutes before Breakfast | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
    0.5 to 1.5 Hours before Breakfast | 165 | 56 | 167 | 52 | 53 | 164 | 50 | 707
    1.5 to 2.5 Hours before Breakfast | 29 | 8 | 35 | 13 | 8 | 27 | 15 | 135
    2.5 to 4 Hours before Breakfast | 5 | 2 | 4 | 3 | 4 | 8 | 1 | 27
Lumbar Spine (L2-L4) Bone Mineral Density (BMD), Categorical [Number; unit: participants] — Data was available for 199, 66, 206, 68, 65, 200 and 66 participants in each treatment arm, respectively. YAM=young adult mean (20 to 44 years age range).
  participants
    Min - ≤0.707 g/cm^2 | 167 | 46 | 176 | 54 | 52 | 158 | 49 | 702
    0.708 (70%YAM) - ≤0.808 g/cm^2 | 24 | 13 | 21 | 11 | 10 | 28 | 11 | 118
    0.809 (80%YAM) g/cm^2 - ≤Max | 8 | 7 | 9 | 3 | 3 | 14 | 6 | 50
L2-L4 (BMD) [Mean (Standard Deviation); unit: g/cm^2] — Data was available for 199, 66, 206, 68, 65, 200 and 66 participants in each treatment arm, respectively.
  g/cm^2 | 0.6553 (0.09060) | 0.6690 (0.11746) | 0.6477 (0.08037) | 0.6633 (0.08766) | 0.6448 (0.08909) | 0.6589 (0.09893) | 0.6714 (0.09999) | 0.6564 (0.09303)
L2-L4 BMD T-score, Categorical [Number; unit: participants] — BMD T-score is a comparison of an individual's BMD compared to "normal". Also, BMD T-score is the standard deviation of the difference between measured BMD and that of the healthy young adult "normal". The T-score scale is as follows: -1 and above=normal, -1 to -2.5=osteopenia (below normal and may lead to osteoporosis), and -2.5 and below=osteoporosis.
  Data was available for 199, 66, 206, 68, 65, 200 and 66 participants in each treatment arm, respectively.
  participants
    Min - ≤-2.500 | 169 | 47 | 177 | 54 | 53 | 160 | 51 | 711
    -2.499 - ≤-1.000 | 28 | 16 | 26 | 12 | 12 | 36 | 12 | 142
    -0.999 - ≤Max | 2 | 3 | 3 | 2 | 0 | 4 | 3 | 17
L2-L4 BMD T-score [Mean (Standard Deviation); unit: score on a scale] — BMD T-score is a comparison of an individual's BMD compared to "normal". Also, BMD T-score is the standard deviation of the difference between measured BMD and that of the healthy young adult "normal". The T-score scale is as follows: -1 and above=normal, -1 to -2.5=osteopenia (below normal and may lead to osteoporosis), and -2.5 and below=osteoporosis. Data was available for 199, 66, 206, 68, 65, 200 and 66 participants in each treatment arm, respectively.
  score on a scale | -2.9889 (0.76130) | -2.8738 (0.98709) | -3.0532 (0.67537) | -2.9219 (0.73670) | -3.0773 (0.74863) | -2.9587 (0.83135) | -2.8536 (0.84030) | -2.9796 (0.78178)
Total Proximal Femur BMD [Mean (Standard Deviation); unit: g/cm^2] — Data was available for 199, 66, 206, 68, 65, 200 and 66 participants in each treatment arm, respectively.
  g/cm^2 | 0.6553 (0.08997) | 0.6573 (0.09537) | 0.6452 (0.08490) | 0.6580 (0.07982) | 0.6486 (0.06973) | 0.6652 (0.08465) | 0.6520 (0.07289) | 0.6548 (0.08464)
Total Proximal Femur BMD T-score [Mean (Standard Deviation); unit: score on a scale] — BMD T-score is a comparison of an individual's BMD compared to "normal". Also, BMD T-score is the standard deviation of the difference between measured BMD and that of the healthy young adult "normal". The T-score scale is as follows: -1 and above=normal, -1 to -2.5=osteopenia (below normal and may lead to osteoporosis), and -2.5 and below=osteoporosis. Data was available for 199, 66, 206, 68, 65, 200 and 66 participants in each treatment arm, respectively.
  score on a scale | -2.1972 (0.89971) | -2.1770 (0.95369) | -2.2982 (0.84903) | -2.1699 (0.79822) | -2.2642 (0.69731) | -2.0978 (0.84652) | -2.2305 (0.72892) | -2.2021 (0.84645)
Trochanter BMD [Mean (Standard Deviation); unit: g/cm^2] — Data was available for 199, 66, 206, 68, 65, 200 and 66 participants in each treatment arm, respectively.
  g/cm^2 | 0.4938 (0.07793) | 0.4954 (0.06803) | 0.4844 (0.06610) | 0.4932 (0.07164) | 0.4879 (0.05653) | 0.5009 (0.06626) | 0.4900 (0.06824) | 0.4925 (0.06914)
Femoral Neck BMD [Mean (Standard Deviation); unit: g/cm^2] — Data was available for 199, 66, 206, 68, 65, 200 and 66 participants in each treatment arm, respectively.
  g/cm^2 | 0.5318 (0.07695) | 0.5258 (0.08147) | 0.5278 (0.07960) | 0.5348 (0.07154) | 0.5245 (0.06293) | 0.5411 (0.08051) | 0.5373 (0.07346) | 0.5327 (0.07712)
Femoral Neck BMD T-score [Mean (Standard Deviation); unit: score on a scale] — BMD T-score is a comparison of an individual's BMD compared to "normal". Also, BMD T-score is the standard deviation of the difference between measured BMD and that of the healthy young adult "normal". The T-score scale is as follows: -1 and above=normal, -1 to -2.5=osteopenia (below normal and may lead to osteoporosis), and -2.5 and below=osteoporosis. Data was available for 199, 66, 206, 68, 65, 200 and 66 participants in each treatment arm, respectively.
  score on a scale | -2.8683 (0.85505) | -2.9358 (0.90523) | -2.9135 (0.88448) | -2.8360 (0.79487) | -2.9501 (0.69920) | -2.7652 (0.89454) | -2.8077 (0.81618) | -2.8594 (0.85690)
Dual-Energy X-Ray Absorptiometry (DXA) Measuring Apparatus [Number; unit: participants]
  QDR-4500 | 14 | 5 | 14 | 5 | 6 | 12 | 6 | 62
  Delphi | 28 | 9 | 29 | 9 | 9 | 26 | 8 | 118
  Discovery | 114 | 38 | 120 | 39 | 35 | 118 | 35 | 499
  Explorer | 43 | 14 | 43 | 15 | 15 | 45 | 17 | 192
Number of Existing Vertebral (Thoracic [Th4] -L4) Fractures [Number; unit: participants] — Data was available for 199, 66, 206, 68, 65, 200 and 66 participants in each treatment arm, respectively.
  participants
    0 | 138 | 32 | 125 | 42 | 38 | 121 | 35 | 531
    1 | 39 | 21 | 61 | 17 | 18 | 58 | 25 | 239
    2 | 12 | 8 | 12 | 7 | 6 | 15 | 6 | 66
    ≥3 | 10 | 5 | 8 | 2 | 3 | 6 | 0 | 34
Fragility Fracture [Number; unit: participants]
  Yes | 86 | 37 | 91 | 32 | 31 | 104 | 36 | 417
  No | 113 | 29 | 115 | 36 | 34 | 97 | 30 | 454
Primary Osteoporosis Diagnosis Criteria 2012 [Number; unit: participants] — Data was available for 199, 66, 206, 67, 65, 201 and 66 participants in each treatment arm, respectively. YAM=young adult mean (lumbar spine: 20 to 44 years age range, proximal femur: 20 to 29 years age range).
  participants
    Fragility Fracture (Vertebrae or Proximal Femur) | 65 | 30 | 82 | 29 | 25 | 80 | 32 | 343
    Fragility Fracture (Other and BMD<YAM*80%) | 21 | 7 | 9 | 3 | 6 | 24 | 4 | 74
    No Fragility Fracture and BMD<=YAM*70% | 113 | 29 | 115 | 35 | 34 | 97 | 30 | 453
Serum 25-hydroxy Vitamin D (25-OH-D), Categorical [Number; unit: participants] — Data was available for 199, 66, 206, 68, 65, 200 and 66 participants in each treatment arm, respectively.
  participants
    Min - ≤14.9 ng/mL | 18 | 8 | 21 | 5 | 8 | 21 | 8 | 89
    15.0 - ≤27.9 ng/mL | 161 | 51 | 157 | 53 | 50 | 160 | 53 | 685
    28.0 ng/mL - ≤Max | 20 | 7 | 28 | 10 | 7 | 19 | 5 | 96
Serum 25-OH-D [Mean (Standard Deviation); unit: ng/mL] — Data was available for 199, 66, 206, 68, 65, 200 and 66 participants in each treatment arm, respectively.
  ng/mL | 21.55 (5.266) | 21.44 (5.423) | 21.46 (5.592) | 21.64 (5.427) | 21.17 (5.248) | 21.52 (5.121) | 20.58 (4.761) | 21.42 (5.288)
Serum C-telopeptide of Type 1 Collagen (CTX) [Mean (Standard Deviation); unit: ng/mL] — Data was available for 199, 66, 205, 68, 65, 200 and 66 participants in each treatment arm, respectively.
  ng/mL | 0.444 (0.1660) | 0.460 (0.1855) | 0.426 (0.1776) | 0.421 (0.1437) | 0.497 (0.1867) | 0.417 (0.1592) | 0.399 (0.1613) | 0.434 (0.1696)
Serum Bone-type Alkaline Phosphatase (BAP) [Mean (Standard Deviation); unit: μg/L] — Data was available for 199, 66, 205, 68, 65, 200 and 66 participants in each treatment arm, respectively.
  μg/L | 15.91 (5.809) | 16.88 (8.617) | 15.83 (6.035) | 15.45 (5.024) | 17.17 (7.354) | 15.13 (5.164) | 15.13 (6.815) | 15.79 (6.142)
Serum Tartrate-resistant Acid Phosphatase 5b (TRACP-5b) [Mean (Standard Deviation); unit: mU/dL] — Data was available for 199, 66, 205, 68, 65, 200 and 66 participants in each treatment arm, respectively.
  mU/dL | 427.1 (154.67) | 424.1 (144.89) | 422.1 (162.07) | 398.4 (127.54) | 444.7 (142.90) | 410.5 (142.09) | 395.0 (128.38) | 418.5 (148.29)
Serum Procollagen 1 N-terminal Peptide (P1NP) [Mean (Standard Deviation); unit: μg/L] — Data was available for 198, 66, 206, 68, 64, 200 and 66 participants in each treatment arm, respectively.
  μg/L | 51.79 (20.357) | 54.91 (27.552) | 50.89 (22.635) | 47.83 (17.120) | 53.43 (22.783) | 48.53 (20.366) | 46.04 (21.714) | 50.44 (21.648)
Urine Type 1 Collagen Cross-linked N-telopeptide (NTX) [Mean (Standard Deviation); unit: nmol BCE/mmol-CRE] — Data was available for 199, 66, 206, 68, 65, 200 and 66 participants in each treatment arm, respectively.
  nmol BCE/mmol-CRE | 56.76 (26.169) | 61.04 (34.808) | 54.98 (23.928) | 53.77 (22.739) | 64.44 (29.535) | 54.48 (23.988) | 53.66 (23.911) | 56.24 (25.871)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Mean Lumbar Spine (L2-L4) Bone Mineral Density (BMD) Measured by Dual Energy X-Ray Absorptiometry (DXA) at End of Study
Description: The change in BMD in the second to the fourth lumbar vertebrae, L2 to L4, and the averages of L2 to L4 at end of study relative to baseline. DXA is a means of measuring BMD through x-ray.
Time Frame: Baseline and End of Study (up to Month 12)
Population: Full Analysis Set (FAS), all randomized participants who received at least 1 dose of study drug, with data available for analyses.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | NE-58095 IR 2.5 mg Once Daily on Awakening | NE-58095 DR 25 mg Once Monthly Following Breakfast | NE-58095 DR 37.5 mg Once Monthly Following Breakfast
Number analyzed (Participants) | 190 | 194 | 181
percent change | 5.07 (4.749) | 3.36 (4.332) | 4.11 (4.654)
Statistical Analysis 1: Comparison: NE-58095 IR 2.5 mg Once Daily on Awakening vs NE-58095 DR 37.5 mg Once Monthly Following Breakfast; Test type: Non-Inferiority or Equivalence — Non-inferiority was tested using t-test at a one-sided significance level of 2.5% and a non-inferiority margin (Δ) of 1.5%; p = 0.1346, t-test, 1 sided; With a non-inferiority margin (Δ) of 1.5%
Statistical Analysis 2: Comparison: NE-58095 IR 2.5 mg Once Daily on Awakening vs NE-58095 DR 25 mg Once Monthly Following Breakfast; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.6711, t-test, 1 sided; With a non-inferiority margin (Δ) of 1.5%
Statistical Analysis 3: Comparison: NE-58095 IR 2.5 mg Once Daily on Awakening vs NE-58095 DR 37.5 mg Once Monthly Following Breakfast; Test type: Superiority or Other; Mean Difference (Final Values) = -0.96, 95% CI 2-sided [-1.920 to 0.001]
Statistical Analysis 4: Comparison: NE-58095 IR 2.5 mg Once Daily on Awakening vs NE-58095 DR 25 mg Once Monthly Following Breakfast; Test type: Superiority or Other; Mean Difference (Final Values) = -1.71, 95% CI 2-sided [-2.617 to -0.794]
Statistical Analysis 5: Comparison: NE-58095 DR 25 mg Once Monthly Following Breakfast vs NE-58095 DR 37.5 mg Once Monthly Following Breakfast; Test type: Superiority or Other; Mean Difference (Final Values) = 0.75, 95% CI 2-sided [-0.166 to 1.658]

2. Secondary Outcome: Percent Change From Baseline in Mean Lumbar Spine (L2-L4) BMD Measured by DXA at Each Visit
Description: The change in BMD in each vertebra, L2 to L4, and the averages of L2 to L4 at each visit relative to baseline. DXA is a means of measuring BMD through x-ray.
Time Frame: Baseline and Month 6, Month 12, and End of Study (Last observation carried forward at Month 12)
Population: FAS, all randomized participants who received at least 1 dose of study drug, with data available for analyses. "n" in the category is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | NE-58095 IR 2.5 mg Once Daily on Awakening | NE-58095 DR 25 mg Once Monthly on Awakening | NE-58095 DR 25 mg Once Monthly Following Breakfast | NE-58095 DR 25 mg Once Monthly 30 Min. After Breakfast | NE-58095 DR 37.5 mg Once Monthly on Awakening | NE-58095 DR 37.5 mg Once Monthly Following Breakfast | NE-58095 DR 37.5 mg Once Monthly 30 Min. After Breakfast
Number analyzed (Participants) | 199 | 66 | 206 | 68 | 65 | 200 | 66
percent change
  Month 6 (n=190, 62, 194, 61, 59, 181, 63) | 3.18 (4.211) | 1.73 (3.635) | 1.92 (4.124) | 2.40 (3.408) | 3.67 (4.841) | 2.70 (4.117) | 2.64 (4.907)
  Month 12 (n=178, 58, 180, 58, 55, 171, 60) | 5.00 (4.783) | 3.83 (4.227) | 3.53 (4.423) | 3.98 (3.784) | 5.04 (4.387) | 4.05 (4.518) | 4.38 (5.277)
  End of Study (n=190, 62, 194, 61, 59, 181, 63) | 5.07 (4.749) | 3.82 (4.158) | 3.36 (4.332) | 3.93 (3.714) | 4.81 (4.383) | 4.11 (4.654) | 4.36 (5.150)

3. Secondary Outcome: Percent Change From Baseline in Femur (Total Proximal Femur) BMD Measured by DXA at Each Visit
Description: The change in BMD in the total proximal femur (whole bone, trochanteric region, and neck region) at each visit relative to baseline. DXA is a means of measuring BMD through x-ray.
Time Frame: Baseline and Month 6, Month 12, and End of Study (Last observation carried forward at Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | NE-58095 IR 2.5 mg Once Daily on Awakening | NE-58095 DR 25 mg Once Monthly on Awakening | NE-58095 DR 25 mg Once Monthly Following Breakfast | NE-58095 DR 25 mg Once Monthly 30 Min. After Breakfast | NE-58095 DR 37.5 mg Once Monthly on Awakening | NE-58095 DR 37.5 mg Once Monthly Following Breakfast | NE-58095 DR 37.5 mg Once Monthly 30 Min. After Breakfast
Number analyzed (Participants) | 199 | 66 | 206 | 68 | 65 | 200 | 66
percent change
  Month 6 (n=189, 62, 194, 61, 59, 180, 63) | 1.10 (2.782) | 0.91 (2.665) | 0.43 (2.666) | 0.54 (2.404) | 0.77 (2.401) | 0.78 (2.420) | 0.55 (2.390)
  Month 12 (n=181, 58, 180, 59, 55, 172, 61) | 2.01 (3.316) | 1.32 (3.399) | 0.95 (3.233) | 1.15 (3.182) | 1.38 (3.013) | 1.45 (2.580) | 1.48 (2.880)
  End of Study (n=189, 62, 194, 61, 59, 180, 63) | 1.96 (3.288) | 1.30 (3.309) | 0.89 (3.172) | 1.15 (3.131) | 1.33 (2.948) | 1.45 (2.565) | 1.39 (2.873)

4. Secondary Outcome: Percent Change From Baseline in Femur (Trochanter) BMD Measured by DXA at Each Visit
Description: The change in BMD in the femur (trochanter) at each visit relative to baseline. DXA is a means of measuring BMD through x-ray.
Time Frame: Baseline and Month 6, Month 12, and End of Study (Last observation carried forward at Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | NE-58095 IR 2.5 mg Once Daily on Awakening | NE-58095 DR 25 mg Once Monthly on Awakening | NE-58095 DR 25 mg Once Monthly Following Breakfast | NE-58095 DR 25 mg Once Monthly 30 Min. After Breakfast | NE-58095 DR 37.5 mg Once Monthly on Awakening | NE-58095 DR 37.5 mg Once Monthly Following Breakfast | NE-58095 DR 37.5 mg Once Monthly 30 Min. After Breakfast
Number analyzed (Participants) | 199 | 66 | 206 | 68 | 65 | 200 | 66
percent change
  Month 6 (n=189, 62, 194, 61, 59, 180, 63) | 1.34 (4.854) | 1.57 (3.832) | 0.70 (4.324) | 0.80 (3.500) | 1.46 (3.495) | 1.09 (3.141) | 0.53 (4.432)
  Month 12 (n=181, 58, 180, 59, 55, 172, 61) | 2.59 (6.007) | 1.80 (4.030) | 1.36 (4.632) | 1.66 (4.095) | 2.47 (4.129) | 1.94 (3.722) | 1.90 (4.259)
  End of Study (n=189, 62, 194, 61, 59, 180, 63) | 2.52 (5.938) | 1.67 (3.951) | 1.35 (4.551) | 1.64 (4.038) | 2.42 (4.005) | 1.94 (3.661) | 1.85 (4.203)

5. Secondary Outcome: Percent Change From Baseline in Femur (Femoral Neck) BMD Measured by DXA at Each Visit
Description: The change in BMD in the femur (femoral neck) at each visit relative to baseline. DXA is a means of measuring BMD through x-ray.
Time Frame: Baseline and Month 6, Month 12, and End of Study (Last observation carried forward at Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | NE-58095 IR 2.5 mg Once Daily on Awakening | NE-58095 DR 25 mg Once Monthly on Awakening | NE-58095 DR 25 mg Once Monthly Following Breakfast | NE-58095 DR 25 mg Once Monthly 30 Min. After Breakfast | NE-58095 DR 37.5 mg Once Monthly on Awakening | NE-58095 DR 37.5 mg Once Monthly Following Breakfast | NE-58095 DR 37.5 mg Once Monthly 30 Min. After Breakfast
Number analyzed (Participants) | 199 | 66 | 206 | 68 | 65 | 200 | 66
percent change
  Month 6 (n=189, 62, 194, 61, 59, 180, 63) | 1.07 (3.406) | 0.90 (3.903) | 0.71 (4.205) | 0.49 (3.804) | 1.01 (3.732) | 0.57 (3.572) | 0.67 (2.770)
  Month 12 (n=181, 58, 180, 59, 55, 172, 61) | 2.00 (4.010) | 0.78 (4.302) | 1.34 (4.687) | 1.47 (4.055) | 1.00 (3.799) | 1.24 (3.492) | 0.56 (4.020)
  End of Study (n=189, 62, 194, 61, 59, 180, 63) | 1.96 (4.017) | 0.99 (4.451) | 1.30 (4.638) | 1.55 (4.009) | 0.96 (3.754) | 1.29 (3.578) | 0.52 (3.962)

6. Secondary Outcome: Percent Change From Baseline in Bone Turnover Marker Serum Creatinine (CTX) at Each Visit
Description: Blood samples for serum bone turnover markers were collected at specified visits according to the study schedule. Blood samples were to be collected at about the same time of the day, as far as possible, throughout the study.
Time Frame: Baseline and Months 1, 3, 6, 9 and 12 and End of Study (Last observation carried forward at Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | NE-58095 IR 2.5 mg Once Daily on Awakening | NE-58095 DR 25 mg Once Monthly on Awakening | NE-58095 DR 25 mg Once Monthly Following Breakfast | NE-58095 DR 25 mg Once Monthly 30 Min. After Breakfast | NE-58095 DR 37.5 mg Once Monthly on Awakening | NE-58095 DR 37.5 mg Once Monthly Following Breakfast | NE-58095 DR 37.5 mg Once Monthly 30 Min. After Breakfast
Number analyzed (Participants) | 199 | 66 | 206 | 68 | 65 | 200 | 66
percent change
  Month 1 (n=199, 66, 204, 68, 65, 200, 66) | -41.02 (27.396) | -17.42 (27.978) | -15.53 (26.107) | -18.80 (25.956) | -33.52 (24.667) | -24.74 (28.675) | -19.34 (28.442)
  Month 3 (n=193, 63, 193, 65, 60, 184, 63) | -47.79 (25.044) | -29.29 (22.794) | -24.80 (31.118) | -28.76 (28.409) | -36.36 (23.925) | -31.30 (28.196) | -29.94 (26.889)
  Month 6 (n=188, 61, 190, 60, 58, 178, 63) | -52.42 (22.926) | -36.97 (29.126) | -24.39 (38.994) | -35.33 (24.539) | -44.28 (24.390) | -37.65 (28.327) | -35.13 (25.910)
  Month 9 (n=185, 60, 185, 59, 55, 175, 61) | -52.44 (26.256) | -33.61 (27.438) | -16.75 (83.047) | -27.99 (32.106) | -42.94 (24.912) | -34.50 (33.805) | -30.97 (32.819)
  Month 12 (n=181, 55, 178, 59, 54, 170, 60) | -48.98 (28.051) | -32.11 (32.662) | -16.42 (64.139) | -23.68 (44.492) | -40.00 (26.613) | -31.56 (36.239) | -24.62 (37.156)
  End of Study (n=199, 66, 204, 68, 65, 200, 66) | -47.61 (28.275) | -29.94 (36.896) | -16.27 (60.895) | -24.33 (43.256) | -39.58 (26.203) | -32.33 (35.959) | -26.28 (36.284)

7. Secondary Outcome: Percent Change From Baseline in Bone Turnover Marker Serum Bone-type Alkaline Phosphatase (BAP) at Each Visit
Description: as for outcome 6
Time Frame: Baseline and Months 1, 3, 6, 9 and 12 and End of Study (Last observation carried forward at Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | NE-58095 IR 2.5 mg Once Daily on Awakening | NE-58095 DR 25 mg Once Monthly on Awakening | NE-58095 DR 25 mg Once Monthly Following Breakfast | NE-58095 DR 25 mg Once Monthly 30 Min. After Breakfast | NE-58095 DR 37.5 mg Once Monthly on Awakening | NE-58095 DR 37.5 mg Once Monthly Following Breakfast | NE-58095 DR 37.5 mg Once Monthly 30 Min. After Breakfast
Number analyzed (Participants) | 199 | 66 | 206 | 68 | 65 | 200 | 66
percent change
  Month 1 (n=199, 66, 205, 68, 65, 200, 66) | -3.04 (11.881) | -2.93 (13.365) | -2.61 (11.351) | -3.61 (12.135) | -4.16 (13.493) | -3.69 (13.142) | -2.44 (10.662)
  Month 3 (n=193, 63, 193, 65, 60, 184, 63) | -21.56 (15.047) | -13.64 (18.499) | -13.31 (17.846) | -15.99 (19.091) | -24.85 (14.835) | -17.52 (18.589) | -13.83 (24.858)
  Month 6 (n=188, 61, 190, 60, 58, 178, 63) | -28.66 (19.087) | -20.92 (23.433) | -17.93 (21.202) | -23.90 (18.990) | -31.06 (14.859) | -24.06 (19.744) | -23.80 (18.352)
  Month 9 (n=185, 61, 185, 59, 55, 175, 61) | -32.84 (17.700) | -25.23 (24.949) | -22.48 (22.233) | -28.00 (20.334) | -33.15 (16.226) | -28.70 (19.536) | -25.84 (21.043)
  Month 12 (n=181, 55, 178, 59, 54, 170, 60) | -34.53 (20.506) | -29.23 (22.721) | -24.91 (21.537) | -30.51 (17.290) | -38.06 (15.153) | -29.58 (21.560) | -27.74 (21.032)
  End of Study (n=199, 66, 205, 68, 65, 200, 66) | -33.34 (21.428) | -26.27 (24.287) | -23.11 (21.553) | -27.21 (19.932) | -33.94 (18.140) | -27.52 (21.962) | -27.08 (21.632)

8. Secondary Outcome: Percent Change From Baseline in Bone Turnover Marker Serum Tartrate-resistant Acid Phosphatase 5b (TRACP-5b) at Each Visit
Description: as for outcome 6
Time Frame: Baseline and Months 1, 3, 6, 9 and 12 and End of Study (Last observation carried forward at Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | NE-58095 IR 2.5 mg Once Daily on Awakening | NE-58095 DR 25 mg Once Monthly on Awakening | NE-58095 DR 25 mg Once Monthly Following Breakfast | NE-58095 DR 25 mg Once Monthly 30 Min. After Breakfast | NE-58095 DR 37.5 mg Once Monthly on Awakening | NE-58095 DR 37.5 mg Once Monthly Following Breakfast | NE-58095 DR 37.5 mg Once Monthly 30 Min. After Breakfast
Number analyzed (Participants) | 199 | 66 | 206 | 68 | 65 | 200 | 66
percent change
  Month 1 (n=199, 66, 205, 68, 65, 200, 66) | -32.38 (17.664) | -17.26 (20.728) | -17.49 (19.406) | -21.05 (17.749) | -30.75 (19.626) | -25.20 (19.726) | -22.06 (20.097)
  Month 3 (n=193, 63, 193, 65, 60, 184, 63) | -37.27 (17.105) | -25.46 (18.567) | -23.85 (22.714) | -27.46 (19.454) | -33.70 (20.735) | -28.36 (20.299) | -27.13 (22.146)
  Month 6 (n=188, 61, 190, 60, 58, 178, 63) | -39.48 (17.702) | -29.15 (21.223) | -23.87 (27.077) | -29.38 (20.340) | -37.16 (18.794) | -31.49 (21.748) | -30.67 (21.385)
  Month 9 (n=185, 61, 185, 59, 55, 175, 61) | -37.64 (19.734) | -25.82 (24.762) | -19.44 (45.595) | -24.78 (22.657) | -32.78 (21.561) | -28.83 (24.971) | -29.71 (23.200)
  Month 12 (n=181, 55, 178, 59, 54, 170, 60) | -34.91 (20.628) | -23.70 (25.425) | -13.25 (63.783) | -20.54 (26.613) | -31.03 (22.287) | -24.31 (26.832) | -23.21 (25.372)
  End of Study (n=199, 66, 205, 68, 65, 200, 66) | -34.76 (20.602) | -22.93 (26.532) | -13.86 (60.015) | -21.29 (26.141) | -31.97 (21.945) | -25.93 (26.283) | -24.46 (25.027)

9. Secondary Outcome: Percent Change From Baseline in Bone Turnover Marker Serum Procollagen 1 N-terminal Peptide (P1NP) at Each Visit
Description: as for outcome 6
Time Frame: Baseline and Months 1, 3, 6, 9 and 12 and End of Study (Last observation carried forward at Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | NE-58095 IR 2.5 mg Once Daily on Awakening | NE-58095 DR 25 mg Once Monthly on Awakening | NE-58095 DR 25 mg Once Monthly Following Breakfast | NE-58095 DR 25 mg Once Monthly 30 Min. After Breakfast | NE-58095 DR 37.5 mg Once Monthly on Awakening | NE-58095 DR 37.5 mg Once Monthly Following Breakfast | NE-58095 DR 37.5 mg Once Monthly 30 Min. After Breakfast
Number analyzed (Participants) | 199 | 66 | 206 | 68 | 65 | 200 | 66
percent change
  Month 1 (n=196, 66, 206, 68, 64, 200, 66) | -6.55 (17.134) | -9.08 (16.765) | -7.70 (15.206) | -9.73 (16.472) | -13.68 (16.892) | -9.86 (14.908) | -10.07 (15.969)
  Month 3 (n=192, 63, 194, 64, 59, 184, 63) | -45.59 (19.379) | -32.19 (27.464) | -29.09 (26.955) | -34.30 (20.730) | -45.91 (22.176) | -36.80 (29.014) | -34.14 (24.153)
  Month 6 (n=187, 61, 191, 60, 57, 178, 63) | -50.83 (22.450) | -39.51 (27.766) | -33.02 (35.354) | -39.21 (23.522) | -51.40 (18.641) | -42.21 (26.918) | -40.90 (26.225)
  Month 9 (n=184, 61, 186, 59, 54, 175, 61) | -46.82 (29.820) | -34.80 (29.523) | -27.74 (38.273) | -36.41 (24.862) | -46.14 (21.531) | -38.32 (30.139) | -32.09 (36.574)
  Month 12 (n=180, 55, 179, 59, 53, 170, 60) | -42.90 (31.614) | -35.65 (27.158) | -25.32 (36.833) | -31.80 (28.472) | -42.75 (24.603) | -31.33 (33.403) | -29.11 (35.904)
  End of Study (n=198, 66, 206, 68, 64, 200, 66) | -41.93 (31.952) | -32.03 (31.584) | -25.51 (35.324) | -30.67 (27.441) | -40.82 (24.646) | -31.74 (31.892) | -29.13 (34.616)

10. Secondary Outcome: Percent Change From Baseline in Bone Turnover Marker Urine Type 1 Collagen Cross-linked N-telopeptide (NTX) at Each Visit
Description: Urine samples for urine bone turnover markers were collected at specified visits according to the study schedule. Urine samples were to be collected at about the same time of the day, as far as possible, throughout the study. Urine NTX was corrected by creatinine value.
Time Frame: Baseline and Months 1, 3, 6, 9 and 12 and End of Study (Last observation carried forward at Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | NE-58095 IR 2.5 mg Once Daily on Awakening | NE-58095 DR 25 mg Once Monthly on Awakening | NE-58095 DR 25 mg Once Monthly Following Breakfast | NE-58095 DR 25 mg Once Monthly 30 Min. After Breakfast | NE-58095 DR 37.5 mg Once Monthly on Awakening | NE-58095 DR 37.5 mg Once Monthly Following Breakfast | NE-58095 DR 37.5 mg Once Monthly 30 Min. After Breakfast
Number analyzed (Participants) | 199 | 66 | 206 | 68 | 65 | 200 | 66
percent change
  Month 1 (n=199, 66, 206, 68, 65, 200, 66) | -32.73 (29.296) | -11.79 (38.228) | -12.42 (35.178) | -17.15 (40.458) | -29.81 (29.087) | -16.42 (39.131) | -12.64 (42.198)
  Month 3 (n=193, 63, 194, 65, 60, 184, 63) | -37.94 (30.360) | -22.32 (35.861) | -15.64 (39.676) | -20.24 (37.412) | -31.27 (28.984) | -22.60 (35.284) | -20.70 (37.137)
  Month 6 (n=188, 61, 191, 60, 58, 178, 63) | -35.00 (35.405) | -29.69 (37.178) | -7.96 (52.202) | -19.51 (41.804) | -36.99 (28.317) | -20.79 (40.913) | -20.92 (38.419)
  Month 9 (n=185, 61, 186, 59, 55, 175, 61) | -30.97 (38.541) | -17.23 (38.383) | -7.71 (50.697) | -19.48 (36.149) | -31.25 (26.172) | -15.90 (47.103) | -14.07 (46.266)
  Month 12 (n=181, 55, 179, 59, 54, 170, 60) | -35.64 (37.715) | -27.45 (33.172) | -4.66 (61.863) | -24.87 (34.422) | -31.74 (34.664) | -17.68 (55.937) | -21.94 (42.649)
  End of Study (n=199, 66, 206, 68, 65, 200, 66) | -35.30 (37.274) | -25.83 (32.786) | -4.72 (59.237) | -23.18 (35.863) | -31.55 (35.083) | -21.06 (53.671) | -24.14 (42.102)

11. Secondary Outcome: Percentage of Participants With New Non-traumatic Vertebral Fractures (Including the Worsening of Pre-existing Fractures)
Description: New non-traumatic vertebral fractures were identified by interpretable X-ray images of 13 vertebrae from the fourth thoracic to the fourth lumbar vertebra. A Central Review Committee member for X-ray determined the presence or absence of new vertebral fractures, the number of new fractures, the presence or absence of worsening pre-existing vertebral fractures, and the number of worsened fractures. The assessment of new vertebral fractures and the worsening of pre-existing vertebral fractures was semiquantitative. The X-ray images were visually inspected and classified into normal (Grade 0), mild deformation (Grade 1), moderate deformation (Grade 2), or severe deformation (Grade 3). If the assessment of any vertebra became worse by at least 1 grade after starting the treatment, its height was measured. A new vertebral fracture or a worsening pre-existing vertebral fracture was concluded if the vertebra's height was reduced from the baseline by at least 20% and by at least 4 mm.
Time Frame: Baseline to Month 12
Population: FAS, all randomized participants who received at least 1 dose of study drug, with data available for analyses.
Measure: Number; unit: percentage of participants
Arm/Group | NE-58095 IR 2.5 mg Once Daily on Awakening | NE-58095 DR 25 mg Once Monthly on Awakening | NE-58095 DR 25 mg Once Monthly Following Breakfast | NE-58095 DR 25 mg Once Monthly 30 Min. After Breakfast | NE-58095 DR 37.5 mg Once Monthly on Awakening | NE-58095 DR 37.5 mg Once Monthly Following Breakfast | NE-58095 DR 37.5 mg Once Monthly 30 Min. After Breakfast
Number analyzed (Participants) | 190 | 61 | 193 | 62 | 59 | 178 | 63
percentage of participants
  Yes | 2.1 | 3.3 | 2.1 | 3.2 | 3.4 | 1.1 | 1.6
  No | 97.9 | 96.7 | 97.9 | 96.8 | 96.6 | 98.9 | 98.4

ADVERSE EVENTS:
Time Frame: First dose of study drug to 30 days past last dose of study drug (Up to 13 Months)
Description: At each visit the investigator documented any occurrence of AEs and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of relation to study treatment. AEs were monitored until the participant recovered or investigator judged no further follow-up was needed.
Arm/Group | NE-58095 IR 2.5 mg Once Daily on Awakening | NE-58095 DR 25 mg Once Monthly on Awakening | NE-58095 DR 25 mg Once Monthly Following Breakfast | NE-58095 DR 25 mg Once Monthly 30 Min. After Breakfast | NE-58095 DR 37.5 mg Once Monthly on Awakening | NE-58095 DR 37.5 mg Once Monthly Following Breakfast | NE-58095 DR 37.5 mg Once Monthly 30 Min. After Breakfast
Serious Adverse Events (participants affected / at risk) | 12/199 | 5/66 | 11/206 | 7/68 | 2/65 | 8/200 | 3/66
Other Adverse Events (participants affected / at risk) | 128/199 | 43/66 | 132/206 | 43/68 | 46/65 | 138/200 | 42/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NE-58095 IR 2.5 mg Once Daily on Awakening (N=199) | NE-58095 DR 25 mg Once Monthly on Awakening (N=66) | NE-58095 DR 25 mg Once Monthly Following Breakfast (N=206) | NE-58095 DR 25 mg Once Monthly 30 Min. After Breakfast (N=68) | NE-58095 DR 37.5 mg Once Monthly on Awakening (N=65) | NE-58095 DR 37.5 mg Once Monthly Following Breakfast (N=200) | NE-58095 DR 37.5 mg Once Monthly 30 Min. After Breakfast (N=66)
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dacryostenosis acquired (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Drowning (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 — One treatment-emergent death occurred during treatment in NE-58095 DR 37.5 mg Once Monthly Following Breakfast group and is not related to study drug.
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Sarcoidosis (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mycobacterial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 0 | 0 | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Brain stem infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NE-58095 IR 2.5 mg Once Daily on Awakening (N=199) | NE-58095 DR 25 mg Once Monthly on Awakening (N=66) | NE-58095 DR 25 mg Once Monthly Following Breakfast (N=206) | NE-58095 DR 25 mg Once Monthly 30 Min. After Breakfast (N=68) | NE-58095 DR 37.5 mg Once Monthly on Awakening (N=65) | NE-58095 DR 37.5 mg Once Monthly Following Breakfast (N=200) | NE-58095 DR 37.5 mg Once Monthly 30 Min. After Breakfast (N=66)
Dry eye (Eye disorders) | 2 | 3 | 3 | 0 | 4 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 9 | 2 | 15 | 8 | 10 | 22 | 3
Constipation (Gastrointestinal disorders) | 10 | 4 | 12 | 2 | 4 | 20 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3 | 14 | 5 | 4 | 15 | 6
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 3 | 2 | 4
Pyrexia (General disorders) | 1 | 1 | 9 | 2 | 3 | 13 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 2 | 4 | 0 | 3 | 1
Nasopharyngitis (Infections and infestations) | 64 | 19 | 51 | 25 | 15 | 42 | 22
Cystitis (Infections and infestations) | 2 | 2 | 8 | 1 | 4 | 10 | 0
Gastroenteritis (Infections and infestations) | 1 | 2 | 5 | 3 | 2 | 10 | 1
Fall (Injury, poisoning and procedural complications) | 21 | 7 | 13 | 3 | 3 | 15 | 5
Contusion (Injury, poisoning and procedural complications) | 16 | 5 | 10 | 1 | 2 | 13 | 7
Ligament sprain (Injury, poisoning and procedural complications) | 8 | 2 | 8 | 0 | 4 | 8 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 5 | 2 | 5 | 1 | 3 | 10 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 14 | 1 | 16 | 5 | 4 | 11 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 13 | 2 | 2 | 13 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 8 | 1 | 4 | 16 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 8 | 3 | 5 | 2 | 4 | 9 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 4 | 0 | 3 | 1
Headache (Nervous system disorders) | 3 | 1 | 10 | 4 | 1 | 5 | 5
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 10 | 5 | 4 | 12 | 2
Eczema (Skin and subcutaneous tissue disorders) | 10 | 3 | 11 | 2 | 3 | 12 | 4
Hypertension (Vascular disorders) | 2 | 1 | 7 | 5 | 2 | 2 | 4

LIMITATIONS AND CAVEATS:
The collaborator company name EA Pharma Co., Ltd. has been changed from 1st April 2016. The legacy name was Ajinomoto Pharmaceutics Co., Ltd.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.